CLINICAL TRIAL: NCT05576610
Title: The Effect of Enzyme-containing Mouth Spray on Oral Health Status and S.Mutans Levels in Paediatric Patients Attending Hospital Universiti Sains Malaysia ( HUSM ) , Kelantan
Brief Title: The Effect of Enzyme-containing Mouth Spray on Oral Health Status and S.Mutans Levels in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ashwini M. Madawana, Principal Investigator, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUSMalaysia
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Gingivitis; Plaque Induced Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enzyme containing mouth spray + Standard Preventive Advice (Experimental): Usage of Oral7 mouth spray along side with the Standard Preventive Advice
  Interventions: Procedure: Standard preventive advice+ enzymatic mouth sprays ( Oral7 mouth spray)
- Normal Saline mouth spray +Standard Preventive Advice (Placebo Comparator): Usage of normal saline containing mouth spray along side with the Standard Preventive Advice
  Interventions: Procedure: Standard Preventive Advice + placebo mouth spray ( normal saline mouth spray )

INTERVENTIONS:
Procedure: Standard preventive advice+ enzymatic mouth sprays ( Oral7 mouth spray) — The following were the advices given face-to-face to parent and participant and a take home pamphlet was provided:
  * Ensure thorough cleaning especially at the gum line and in the areas between the teeth.
  * To not share toothbrushes.
  * To use toothpaste containing fluoride at least 1000ppm fluoride concentration.
  * To store toothbrushes apart to prevent spread of diseases through the bristles.
  * To brush teeth at least twice a day, after meals and before bed.
  * To brush for as long as two to three minutes.
  * Parents would be advised told to supervise the participant's brushing.
  Frequency of using the Mouth spray would be two puffs, three times a day that is in the morning after waking up, during tea time and before sleep. A squirt is to be applied to the right/left side of the mouth on the buccal aspect and a squirt on the lingual aspect. Parents will be asked to apply the spray and to supervise children during oral hygiene procedures.
  Other Names: Oral7 mouth spray
  Arms: Enzyme containing mouth spray + Standard Preventive Advice
Procedure: Standard Preventive Advice + placebo mouth spray ( normal saline mouth spray ) — The following were the advices given face-to-face to parent and participant and a take home pamphlet was provided:
  * Ensure thorough cleaning especially at the gum line and in the areas between the teeth.
  * To not share toothbrushes.
  * To use toothpaste containing fluoride at least 1000ppm fluoride concentration.
  * To store toothbrushes apart to prevent spread of diseases through the bristles.
  * To brush teeth at least twice a day, after meals and before bed.
  * To brush for as long as two to three minutes.
  * Parents would be advised told to supervise the participant's brushing.
  Frequency of using the mouth spray would be two puffs, three times a day that is in the morning after waking up, during tea time and before sleep. A squirt is to be applied to the right/left side of the mouth on the buccal aspect and a squirt on the lingual aspect. Parents will be asked to apply the spray and to supervise children during oral hygiene procedures.
  Other Names: Normal Saline Mouth Spray
  Arms: Normal Saline mouth spray +Standard Preventive Advice

SUMMARY:
An interventional study was done on evaluating the Effect of Enzyme-containing Mouth Spray on Oral Health Status and S.Mutans levels in Paediatric Patients attending Hospital Universiti Sains Malaysia ( HUSM ) , Kelantan. This study compared the gingivitis score , plaque score and saliva bacteria count between the patients receiving a standard preventive advice alongside with normal saline mouth spray and those receiving standard preventive advice alongside with an enzyme containing mouth spray .

DETAILED DESCRIPTION:
General Objective

To evaluate the effect of enzyme-containing mouth sprays on children's oral health compared to those receiving normal saline mouth spray with standard preventive advice after a 4-week follow-up.

Specific Objectives

1. To compare the mean plaque score in children using enzyme-containing mouth sprays with standard preventive advice compared to children receiving normal saline mouth spray with standard preventive advice after a 4-week follow-up.
2. To compare the mean gingivitis score in children using enzyme-containing mouth sprays with standard preventive advice compared to children receiving normal saline mouth spray with standard preventive advice after a 4-week follow-up.
3. To compare the mean saliva bacterial count in children using enzyme-containing mouth sprays with standard preventive advice compared to children receiving receiving normal saline mouth spray with standard preventive advice after a 4-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children of age group 4-7

Exclusion Criteria:

* Children with medical problems
* Children with Special Needs
* Uncooperative Children ( Level of Cooperation would be measured using Frankl's behavior scale)

Reviewer's comment : To list down Frankl's Classification and how we define uncooperative

As per AAPD 2022 , The Frankl behavior rating scale is a frequently used behavior rating systems in both clinical dentistry and research. This scale indicates observed child's behaviors into four categories (1; Definitely negative, 2; Negative, 3; Positive, 4; Definitely positive)

1. _ _ Definitely negative. Refusal of treatment, forceful crying, fearfulness, or any other overt evidence of extreme negativism.
2. _ Negative. Reluctance to accept treatment, uncooperative, some evidence of negative attitude but not pronounced (sullen, withdrawn).
3. + Positive. Acceptance of treatmen, cautious behavior at times, willingness to comply with the dentist, at times with reservation, but patient follows the dentist's directions cooperatively.
4. ++ Definitely positive. Good rapport with the dentist, interest in the dental procedures, laughter and enjoyment

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Plaque Score | 4 weeks
  Was measured using the Silness-Loe Plaque Index 1964 from each patient before and after the intervention in both control and case study groups and the mean score and standard deviation was recorded in a table.
  Scoring Criteria 0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth.
  2. Moderate accumulation of deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  PIaque Score formula:
  Total scores / No of teeth examined
  Range of scores :
  Excellent : 0 Good : 0.1-0.9 Fair: 1.0-1.9 Poor: 2.0-3.0

SECONDARY OUTCOMES:
Gingivitis Score | 4 weeks
  Was measured using the Loe and Silness Gingival Index 1963 from each patient before and after the intervention in both control and case study groups and the mean score and standard deviation would be recorded in a table.
  Scoring Criteria 0 No inflammation.
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
  Gingivitis score for the individual would be calculated using a formula as follows :
  Sum of indices of teeth / no of teeth examined
  These scores was then classified into either a Mild , Moderate or Severe form of Gingivitis as follows :
  Mild gingivitis : 0.1-1.0 Moderate gingivitis : 1.1-2.0 Severe gingivitis : 2.1-3.0

OTHER OUTCOMES:
Saliva Bacterial Count | 4 weeks
  The saliva sample was collected from 3 patients each of both case control and study groups before and after the intervention. Saliva samples were collected at the start of the study that is during the delivery of the short dental hygiene educational message, and after 4 weeks. Every child involved was then told to spit in a centrifuge tube to obtain 1-2 ml of total volume. The saliva was then cultured in the lab for saliva bacteria analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ashwini M.Madawana, BDS, Principal Investigator — Hospital Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual Participant data would be protected under the Ethical Board of Hospital University Sains Malaysia .